CLINICAL TRIAL: NCT02366078
Title: The Efficacy of Using Blended Learning With the Stress Management and Resilience Training (SMART) Program to Decrease Stress and Enhance Resilience in Public School Staff
Brief Title: Stress Management Training for School Staff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brent A. Bauer, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14-005976
Record Dates: First submitted 2015-02-11; First posted 2015-02-19 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stress management (Experimental): Participants will receive SMART traiing
  Interventions: Behavioral: SMART

INTERVENTIONS:
Behavioral: SMART — Paced breathing meditation with cognitive training

SUMMARY:
The purpose of this study is to investigate the outcomes of the Stress Management and Resiliency Training (SMART) program among Public School staff in 2 communities in Minnesota. Feasibility of a blended in-person and online teaching approach of the program will also be evaluated.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the outcomes of the Stress Management and Resiliency Training (SMART) program among Public School staff in 2 communities in Minnesota. Feasibility of a blended in-person and online teaching approach of the program will also be evaluated.

This study builds on previous work in other working populations with high stress levels inherent in the specific work process.

ELIGIBILITY:
Inclusion Criteria:

* Public school teacher
* Able tor read English

Exclusion Criteria:

* Unable to read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Self reported stress level | 1 year
  Linear analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Brent Bauer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No